CLINICAL TRIAL: NCT06458855
Title: Pilot Trial: Pilot Study of Somatic-Autonomic Nerve Grafting Technique to Restore Erectile Function in Patients With Persistent Erectile Dysfunction Post Radical Prostatectomy
Brief Title: Nerve Grafting Technique to Restore Erectile Function Post Radical Prostatectomy
Acronym: PRP-NR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Victor McPherson, MD, MSc, FRCSC, Assistant Professor Division of Urology, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-4130
Record Dates: First submitted 2024-05-21; First posted 2024-06-14 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer; Erectile Dysfunction Following Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PRP-NR (Experimental): Post radical prostatectomy nerve restoration procedure
  Interventions: Procedure: Post radical prostatectomy nerve restoration procedure (PRP-NR)

INTERVENTIONS:
Procedure: Post radical prostatectomy nerve restoration procedure (PRP-NR) — A somatic to autonomic nerve grafting procedure which will use a nerve graft of ilioinguinal nerve harvested from the inguinal canal to perform a bilateral end to side junction between the dorsal penile nerve and the penile corpora cavernosa

SUMMARY:
A single arm prospective pilot trial evaluating the safety and the 1-year erectile recovery outcomes of patients undergoing a somatic to autonomic nerve grafting procedure for restoration of erectile function in patients who have lost erectile function following radical prostatectomy for prostate cancer. During this study a total of 10 patients who have persistent erectile dysfunction for more than 18 months post prostatectomy will undergo a post radical prostatectomy nerve restoration procedure (PRP-NR).

DETAILED DESCRIPTION:
The investigators are proposing a single arm prospective pilot study evaluating the safety and the 1-year erectile recovery outcomes of patients undergoing the PRP-NR procedure. A total of 10 patients will undergo the PRP-NR procedure, which is a novel nerve grafting procedure which will utilize a graft of the ilioinguial nerve to perform a bilateral end to side connection between the dorsal penile nerve and the corpora cavernosa with the intent to restore erectile function. Participants will have a baseline evaluation with IIEF-5 and SF-MPQ questionnaires, and then will have re-evaluation with these questionnaires at their standard of care post operative visits at 4 weeks, 3-, 6-, 12-, 18- and 24- months. Post operative safety will be assessed by recording any clinically detected complications during their peri- and post-operative care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with persistent post prostatectomy erectile dysfunction more than 18 months from prostatectomy and which results in the inability to achieve intercourse with the aid of PDE5-I medications.
2. Patients must have had good pre-prostatectomy erectile function with a baseline IIEF score of ≥17 on self-reported assessment of historic function.

Exclusion Criteria:

1. Patients with previous pelvic radiotherapy
2. Patients aged < 18 years at diagnosis
3. Legally incapable patients
4. Patients who are unable to complete questionnaires and have no companion to help complete them
5. Patients with pre-existing neurologic disease
6. Patients with a history of bilateral surgeries for inguinal hernia repair.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is specifically the safety of the operation. This will be measured by adverse events as defined by the Clavian-Dindo classification.The measurement varies from Grade I (Best possible outcome) to Grade V (Worst possible outcome). | Through study completion, an average of 2 years
  Grade I - Deviation from normal p/o course. No pharmacological or surgical treatment, endoscopic or radiological interventions were required. Acceptable therapeutic drugs such as anti-emetics, antipyretics, analgesics, diuretics,electrolytes, physiotherapy. Wound infections, small abscess requiring incision at bedside.
  Grade II - Normal course altered. Pharmacological management other than in Grade I. Blood transfusions and total parenteral nutrition are also included.
  Grade III - Complications that require intervention of various degrees. Grade IIIa are complications that require an intervention performed under local anaesthesia. Grade IIIb are interventions that require general or epidural anaesthesia.
  Grade IV - Complications threatening life of patients (including Central Nervous System complications), requiring Intensive Treatment Unit support. Grade IVa are single organ dysfunction (including dialysis). Grade IVb is multi-organ dysfunction.
  Grade V - Death of a patient.

SECONDARY OUTCOMES:
International Index of Erectile Function-5 (IIEF-5) | 4 weeks post PRP-NR
  The IIEF-5 is used to determine the prevalence of erectile dysfunction (ED) in a non-selected population using the abridged 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool.
  Each answer has a score from 1 (very low) to 5 (very high). The sum of all the answers gives a final result of 1-7 (Severe ED - Worst Outcome), 8-11 (Moderate ED), 12-16 (Mild-moderate ED), 17-21 (Mild ED) and 22-25 (No ED - Best Outcome).
International Index of Erectile Function-5 (IIEF-5) | 3 months post PRP-NR
  The IIEF-5 is used to determine the prevalence of erectile dysfunction (ED) in a non-selected population using the abridged 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool.
  Each answer has a score from 1 (very low) to 5 (very high). The sum of all the answers gives a final result of 1-7 (Severe ED - Worst Outcome), 8-11 (Moderate ED), 12-16 (Mild-moderate ED), 17-21 (Mild ED) and 22-25 (No ED - Best Outcome).
International Index of Erectile Function-5 (IIEF-5) | 6 months post PRP-NR
  The IIEF-5 is used to determine the prevalence of erectile dysfunction (ED) in a non-selected population using the abridged 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool.
  Each answer has a score from 1 (very low) to 5 (very high). The sum of all the answers gives a final result of 1-7 (Severe ED - Worst Outcome), 8-11 (Moderate ED), 12-16 (Mild-moderate ED), 17-21 (Mild ED) and 22-25 (No ED - Best Outcome).
International Index of Erectile Function-5 (IIEF-5) | 12 months post PRP-NR
  The IIEF-5 is used to determine the prevalence of erectile dysfunction (ED) in a non-selected population using the abridged 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool.
  Each answer has a score from 1 (very low) to 5 (very high). The sum of all the answers gives a final result of 1-7 (Severe ED - Worst Outcome), 8-11 (Moderate ED), 12-16 (Mild-moderate ED), 17-21 (Mild ED) and 22-25 (No ED - Best Outcome).
International Index of Erectile Function-5 (IIEF-5) | 18 months post PRP-NR
  The IIEF-5 is used to determine the prevalence of erectile dysfunction (ED) in a non-selected population using the abridged 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool.
  Each answer has a score from 1 (very low) to 5 (very high). The sum of all the answers gives a final result of 1-7 (Severe ED - Worst Outcome), 8-11 (Moderate ED), 12-16 (Mild-moderate ED), 17-21 (Mild ED) and 22-25 (No ED - Best Outcome).
International Index of Erectile Function-5 (IIEF-5) | 24 months post PRP-NR
  The IIEF-5 is used to determine the prevalence of erectile dysfunction (ED) in a non-selected population using the abridged 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool.
  Each answer has a score from 1 (very low) to 5 (very high). The sum of all the answers gives a final result of 1-7 (Severe ED - Worst Outcome), 8-11 (Moderate ED), 12-16 (Mild-moderate ED), 17-21 (Mild ED) and 22-25 (No ED - Best Outcome).
Short Form McGill Pain Questionnaire (SF-MPQ) | 4 weeks post PRP-NR
  The SF-MPQ was designed to measure post-surgical pain. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors.
  The sum of the scores gives a range of outcomes; a score of 0 (no pain - Best Possible Outcome) to a score of 45 (Most severe pain - Worst Possible Outcome)
Short Form McGill Pain Questionnaire (SF-MPQ) | 3 months post PRP-NR
  The SF-MPQ was designed to measure post-surgical pain. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors.
  The sum of the scores gives a range of outcomes; a score of 0 (no pain - Best Possible Outcome) to a score of 45 (Most severe pain - Worst Possible Outcome)
Short Form McGill Pain Questionnaire (SF-MPQ) | 6 months post PRP-NR
  The SF-MPQ was designed to measure post-surgical pain. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors.
  The sum of the scores gives a range of outcomes; a score of 0 (no pain - Best Possible Outcome) to a score of 45 (Most severe pain - Worst Possible Outcome)
Short Form McGill Pain Questionnaire (SF-MPQ) | 12 months post PRP-NR
  The SF-MPQ was designed to measure post-surgical pain. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors.
  The sum of the scores gives a range of outcomes; a score of 0 (no pain - Best Possible Outcome) to a score of 45 (Most severe pain - Worst Possible Outcome)
Short Form McGill Pain Questionnaire (SF-MPQ) | 18 months post PRP-NR
  The SF-MPQ was designed to measure post-surgical pain. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors.
  The sum of the scores gives a range of outcomes; a score of 0 (no pain - Best Possible Outcome) to a score of 45 (Most severe pain - Worst Possible Outcome)
Short Form McGill Pain Questionnaire (SF-MPQ) | 24 months post PRP-NR
  The SF-MPQ was designed to measure post-surgical pain. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors.
  The sum of the scores gives a range of outcomes; a score of 0 (no pain - Best Possible Outcome) to a score of 45 (Most severe pain - Worst Possible Outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Victor McPherson, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada